CLINICAL TRIAL: NCT06002178
Title: Ultrasound Evaluation of the Vascular Anatomy of the Neck to Minimize the Accidental Risk of Vascular Puncture During Percutaneous Tracheostomy
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Principal Investigator, University of Padova
Other Study IDs: AOP3019/2023
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Tracheostomy Complication; Trachea
MeSH Terms: conditions — Tracheal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing surgical procedure: The following variables will be collected: age, weight, height, gender, previous neck surgery/radiotherapy, previous tracheostomy.
  Subsequently, through ultrasound examination, the vascular anatomy of the neck will be studied by dividing it into twelve anatomical quadrants: Four medial quadrants (thyroid membrane, cricoid membrane, and cricothyroid membrane; first tracheal ring, from the beginning of the second tracheal ring to the end of the third tracheal ring), laterally on both right and left sides of each quadrant, the lateral quadrants will be identified. An ultrasound examination with a linear probe with doppler technique will be performed for each quadrant to identify the vascular structures.
  For each quadrant, the presence of vessels, arterial or venous nature, and their diameter will be collected.
  Interventions: Diagnostic Test: Neck ultrasound

INTERVENTIONS:
Diagnostic Test: Neck ultrasound — A neck ultrasound will be performed in order to map superficial arteries and veins of the neck

SUMMARY:
Tracheostomy is a commonly performed procedure in Intensive Care and its incidence tends to increase over time as a consequence of the increase in chronic diseases and the average age of the population accessing Intensive Care.

Surgical open tracheostomy (ST) is the standard procedure but has a relatively high incidence of peristomal infections and perioperative bleeding. Percutaneous dilatational tracheostomy (PDT) was introduced in 1985 and has since become a common bedside procedure. Compared to open ST, PDT has the advantages of a lower risk of wound infection, lower bleeding-related mortality, shorter procedure times, and improved cost-effectiveness.

Fiberoptic bronchoscopy is commonly used during PDT to verify the safety of direct tracheal access [5]. However, bronchoscopy-guided PDT has several limitations regarding the precise identification of cervical anatomical structures and the prevention of complications such as vascular injury.

Preliminary ultrasound examination of neck anatomy has numerous potential benefits, including increased safety during the procedure, identification of cervical vascularization, and localization of the tracheal puncture site with lower risk of complications [6-8]. Several studies have shown that the use of ultrasound in a preliminary and real-time manner can improve first-pass success rate and puncture accuracy, reduce procedure time, and complications.

The objective of this study is to map the arterial and venous vascular anatomy of the neck in order to identify points with a lower risk of vascular injury during PDT. This helps prevent bleeding during tracheostomy, which is one of the major complications associated with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients of eighteen years or older
* Informed consent

Exclusion Criteria:

* Tracheostomized patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients accessing the operating room for any reason
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Mapping of artery and veins of the neck in the general population | through study completion, an average of 1 year
  Described as the size of veins and arteries in the neck
Size of artery and veins of the neck in the general population | through study completion, an average of 1 year
  Described as the size of veins and arteries in the neck

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Padova, Padua, Veneto, Italy

IPD SHARING:
Plan to Share IPD: Undecided